CLINICAL TRIAL: NCT01318200
Title: International Randomized Study of Transarterial Chemoembolization Versus CyberKnife® for Recurrent Hepatocellular Carcinoma
Brief Title: Transarterial Chemoembolization (TACE) vs. CyberKnife for Recurrent Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Accuray Incorporated (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCH001.0
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: Primary liver cancer; Hepatocellular carcinoma; CyberKnife; Accuray; TACE; Transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transarterial Chemoembolization (Active Comparator)
  Interventions: Procedure: Transarterial Chemoembolization
- CyberKnife SBRT (Active Comparator)
  Interventions: Radiation: CyberKnife SBRT

INTERVENTIONS:
Procedure: Transarterial Chemoembolization — Transarterial Chemoembolization will be given within 12 weeks and up to 3 staged procedures, depending on the architecture of the tumor vasculature.
  Arms: Transarterial Chemoembolization
Radiation: CyberKnife SBRT — Dose is 45 Gy (15 Gy in 3 fractions) or 36 Gy(12 Gy in 3 fractions). Tumors should receive the higher dose unless normal tissue constraints cannot be met.
  Arms: CyberKnife SBRT

SUMMARY:
To compare the efficacy of Transarterial Chemoembolization (TACE) to CyberKnife stereotactic body radiotherapy in the treatment of patients with locally recurrent hepatocellular carcinoma (HCC) after TACE.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third most deadly cancer in the world. It is primarily seen in areas where hepatitis is endemic, such as Asia, but other risk factors include alcoholic cirrhosis.

Surgical resection and/or transplantation remain the only curative options. However, more than 80% of patients present with unresectable disease. For these patients with unresectable tumors, a variety of treatment options are available, including transarterial chemoembolization (TACE), radiofrequency ablation (RFA), radioactive microspheres, microwave coagulation, laser-induced thermotherapy, and percutaneous alcohol injection, all of which have similar survival rates. Stereotactic body radiotherapy (SBRT) for unresectable HCC is a relatively new treatment option made available because of significant improvements in diagnostic imaging and radiation delivery techniques. Although follow-up is limited, results show encouraging local control rates. Some investigators have combined TACE with fractionated conventional radiotherapy as a means of intensifying local therapy, with evidence of efficacy.

TACE remains the dominant mode of local therapy for unresectable HCC. However, recurrence rates are high. Because SBRT is rapidly becoming an accepted local therapy for hepatic lesions, its role in treating HCC needs to be further defined. Moreover, once patients have recurred after initial TACE, it is unclear if additional TACE will be as effective or if another mode of local therapy such as SBRT would be preferable.

We propose to conduct a multicenter randomized study comparing TACE vs. SBRT using CyberKnife for locally recurrent HCC. Locally recurrent HCC will include lesions that persist, progress or recur minimum 3 months after initial TACE.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hepatocellular carcinoma by one of the following:

  1. Histopathology
  2. One radiographic technique that confirms a lesion >2 cm with arterial enhancement with washout on delayed phase.
* Hepatic lesion in patients for whom surgical resection is not possible or would not result in an opportunity for cure.
* Radiographic evidence of persistent, progressive or recurrent disease in an area previously treated with TACE. This evaluation should be determined after 6 weeks of initial TACE.
* Multi-specialty evaluation whereby the recurrent liver lesion was deemed by both the attending radiation oncologist and interventional radiologist amenable to treatment by the respective modality

  1. Eligible patients must undergo an IV contrast CT scan of the liver within 6 weeks of enrollment onto the study; a contrast enhanced liver MRI may be substituted for the contrast liver CT
  2. A recent serum AFP must be obtained within 4 weeks of enrollment.
* Unifocal liver tumors not to exceed 7.5 cm in greatest axial dimension. Multifocal lesions will be restricted to lesions that can be treated within a single target volume within the same liver segment and to an aggregate of 7.5 cm as long as the dose constraints to normal tissue can be met.
* Eastern Clinical Oncology Group performance status 0, 1 or 2 (Appendix I).
* Patients with liver disease classified as Child Pugh class A/B, if Child's class B, score must be 8 or less.
* Life expectancy >= 6 months
* Age >= 18 years old
* Albumin >= 2.5 g/dL
* Total Bilirubin <= 3 mg/dL
* INR <= 1.5
* Creatinine <= 2.0 mg/dL
* Both men and women and members of all races and ethnic groups are eligible for this study
* Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation for the recurrent liver tumor
* Prior radiotherapy to the upper abdomen
* Prior RFA to index lesion
* Liver transplant
* Tumors greater than 7.5 cm in greatest axial dimension
* Portal vein thrombus
* Large varices within 2 cm of index lesion (seen on cross section imaging)
* Contraindication to receiving radiotherapy
* Active gastrointestinal bleed within 2 weeks of study enrollment
* Ascites refractory to medical therapy
* Women who are pregnant
* Administration of chemotherapy within the last 1 month
* Presence of multifocal lesions located in different lobes of the liver or extrahepatic metastases
* Participation in another concurrent systemic treatment protocol
* Prior history of malignancy other than HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Freedom from local progression | 12 months
  Freedom from local progression at time T is defined as lack of local progression in the treated liver lesion in the set of patients alive and on study at time T and without distant progression up to time T.

SECONDARY OUTCOMES:
Progression-free survival | 6, 12 and 18 months
  Progression-free survival will be defined as subject alive and free from local progression, disease recurrence elsewhere in the liver, extrahepatic progression, or clinical deterioration unattributable to another underlying medical condition in the absence of clear radiographic findings of progressive disease.
Overall survival | Up to three years following therapy
  Overall survival will be determined as a measure of time from diagnosis of initial recurrence until death from any cause.
Serum AFP levels | 3, 6, 12 and 18 months
  Serum AFP levels will be measured at specific points during the study. The 2 endpoints to be analyzed are:
  * Initial AFP levels
  * AFP response - the percent decrease in serum AFP levels from the initial result to the eventual nadir after therapy
  These endpoints will be correlated to the clinical endpoints (freedom from local progression, progression free-survival, and overall survival).
Freedom from local progression | 6 and 18 months
  Freedom from local progression at time T is defined as lack of local progression in the treated liver lesion in the set of patients alive and on study at time T and without distant progression up to time T.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, MD, PhD, Study Chair — Stanford Comprehensive Cancer Center; Daniel Chang, MD, Study Chair — Stanford Comprehensive Cancer Center; Nishita Kothary, MD, Study Chair — Stanford Comprehensive Cancer Center
Locations (1):
- Stanford Comprehensive Cancer Center, Stanford, California, United States

REFERENCES:
- See also: Information on CyberKnife — http://www.cyberknife.com
- See also: Sponsor website — http://www.accuray.com